CLINICAL TRIAL: NCT06750679
Title: The Effect of Manual Lymph Drainage Applied As an Adjunct to Compression Therapy on Edema and Fibrosis in Individuals with Lower Extremity Lymphedema: a Single Blinded Randomized Controlled Trial
Brief Title: The Effect of Manual Lymph Drainage Applied As an Adjunct to Compression Therapy on Edema Lower Extremity Lymphedema:
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Elif Duygu, assistant professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAIBU-FTR-ED-004
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Lower Extremity Lymphedema
Keywords: lower extremity lymphedema; fibrosis; manual lymphatic drainage; Complex decongestive physiotherapy; Quality of life
MeSH Terms: conditions — Fibrosis | interventions — Compression Bandages

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compression Group (Active Comparator): In compression therapy, multicomponent inelastic compression bandages bandages will be applied (Misra et al., 2023). The individual will be fitted with a stockinet beforehand. Fingers will be bandaged. Then, the extremity will be cylindricalized with a cotton roller or sponge. Subsequently, the foot and ankle will be bandaged using a 6 cm short-stretch bandage. An 8 cm short-stretch bandage will be applied starting from the foot and progressing upward above the ankle. A 10 cm short-stretch bandage will then be applied, beginning at the ankle and wrapping upward. The next bandages will be wrapped upwards starting from the places where the pressure is low. The compression bandage will remain on the patient's leg for approximately 23 hours. When the individual arrives the next day, the bandage will be removed and reapplied. The application time of the inelastic bandage is approximately 20-30 minutes. Compression therapy will be applied 5 days a week for 4 weeks (20 sessions)
  Interventions: Other: Compression bandage
- Compression+MLD Group (Experimental): Participants in the group receiving MLD in addition to compression therapy will undergo a 30-40-minute MLD session to facilitate the entry of interstitial fluid into lymphatic capillaries and enhance lymph propulsion (Misra et al., 2023). The MLD will be performed with gentle pressure of approximately 30-40 mmHg, ensuring the skin and connective tissue move together without sliding on the skin.
  After the MLD session, a multilayer bandaging will be applied to the extremity, which the patient will wear for approximately 23 hours. The bandage will be removed and reapplied during the patient's visit the following day.
  The combined therapy of compression and MLD will be administered five days a week for four weeks (20 sessions in total). Each session will last approximately 50-70 minutes.
  Interventions: Other: Manual lymphatic drainage added to compression

INTERVENTIONS:
Other: Compression bandage — A multicomponent inelastic compression bandage will be applied to the patient. Skin care and simple exercises will be added to intervention
  Arms: Compression Group
Other: Manual lymphatic drainage added to compression — Manual lymphatic drainage will be added to multicomponent inelastik compression bandage, skin care and simple exercises
  Arms: Compression+MLD Group

SUMMARY:
Lymphedema is much more than a disease with edema. Impaired lymphatic drainage triggers adipose tissue deposition and fibrosis. Fibrosis causes lymphatic vessel dysfunction. Therefore, treatment of fibrosis is important. The gold standard of treatment for lymphedema is complex decongestive physiotherapy. In this treatment method consisting of two phases and four components in each phase, each component has its own effect. Compression is the main component of these components in terms of edema reduction. The effect of manual lymph drainage, another component, on edema and fibrosis is contradictory. Although there are studies evaluating fibrosis in lower extremity lymphedema in the literature, there is no study evaluating the effect of treatment on fibrosis and comparing two different methods evaluating fibrosis.

Research question: What is the effect of manual lymph drainage in addition to compression therapy on fibrosis, edema, skin and subcutaneous tissue thickness, and quality of life.

The primary aim of this study was to evaluate the effect of manual lymph drainage applied as an adjunct to compression therapy on fibrosis in individuals with lower extremity lymphedema. The secondary aim of the study was to evaluate the effect of manual lymph drainage in addition to compression therapy on skin and subcutaneous tissue thickness, edema and quality of life.

Patients with lower extremity lymphedema will be randomly allocated to the compression group and manual lymph drainage + compression group. Fibrosis in the tissues of the individuals will be evaluated by ultrasound and SkinFibrometer device, skin and subcutaneous tissue thickness will be evaluated by ultrasound, edema perimeter measurement will be converted to volume, and quality of life will be evaluated by Lymphedema Quality of Life Questionnaire-Lower Extremity before and after treatment. Individuals will be randomized to either 20 sessions of compression bandage or 20 sessions of compression bandage with manual lymph drainage. Both groups will include skin care and exercise components of complex decongestive physiotherapy.

This study will provide important data on whether manual lymph drainage is clinically necessary in the treatment of lower limb lymphedema.

DETAILED DESCRIPTION:
Lower extremity lymphedema (LE) is a chronic disease characterized by the accumulation of protein-rich fluid in the interstitial space and inflammation. It is classified as primary and secondary lymphedema. Primary LE is caused by developmental defects of the lymphatic system, whereas secondary LE is caused by subsequent damage to the lymphatic system. The biggest cause of secondary LE in western countries is cancer surgery.

Lower extremity LE is not a disease characterized only by edema. As the disease progresses, adipose tissue increases and fibrosis is observed. Fibrosis is defined as excessive accumulation of extracellular matrix products. Fibrosis is a well-known cause of organ dysfunction in many systems, including the liver, kidney, heart, and skin. This condition also occurs in limb LL and is a characteristic pathological change seen in LL. The increase in adipose tissue and fibrosis triggered by the presence of lymph fluid leads to increased skin and subcutaneous tissue thickness. These changes increase as the duration and stage of the disease progress.

Inflammation due to impaired lymph drainage triggers the fibrosis process. Histological and immunohistochemical specimens from clinical and experimental skin tissues of patients with LE reveal an increase in collagen fibers in edematous skin due to fibrosis. Fibrosis in LE is not limited to the skin but has also been detected in subcutaneous tissue, including adipose tissue. It has been reported that adipocytes in adipose tissue with LE have hypertrophic changes and larger adipose tissue lobules, and these lobules are surrounded by thick collagen fibers and interstitial lymphatic fluid. It has been reported that collagen accumulation in subcutaneous fat was observed in mouse models of LE. This leads to hardening of the tissue , resulting in non-depressed edema. Fibrosis in the tissue causes lymphatic vessel dysfunction and reduces lymphatic capacity, leading to worsening of LE. It has been reported that fibrotic changes in lymphedema can be partially reversed with complex decongestive physiotherapy (CDF). CDF is a conservative treatment method accepted as the gold standard in the treatment of LE. It consists of two phases: discharge and protection. While the unloading phase aims to reduce limb volume, the preservation phase aims to maintain the reduced volume. The unloading phase consists of 4 main components: manual lymph drainage (MLD), skin care, compression, and exercise. In the protection phase, compression bandages are replaced by compression garments, and manual lymph drainage is replaced by self/simple lymph drainage. The drainage phase lasts at least 2-4 weeks, and the protection phase lasts for life Each treatment component has a unique mechanism of action in the treatment of lymphedema. MLD is a gentle massage technique that aims to move the skin and connective tissue, thus stretching the anchor filaments connected to the lymphatic capillaries and opening the lymphatic capillaries without causing hyperemia. There are different holding techniques. MLD is thought to increase the transport rate of lymphatic fluid, develop new pathways for lymphatic drainage from edematous areas to adjacent non-edematous areas, remove protein deposits from the tissue, and break down fibrotic tissue. Compression is to create more tissue pressure during contractions by resisting muscle activity. This is the strongest stimulation for lymph drainage. Compression also prevents fluid accumulation in the tissue by reducing capillary filtration. It allows resorption of fluid in the interstitial space. It displaces fluid to non-compressed areas where drainage is normal. Compression is also thought to be effective in the destruction of fibrosclerotic tissue.

In the literature, the effect of MLD and compression applications on edema has been frequently evaluated, and the effectiveness of compression bandaging has been shown, although the effect of MLD on edema reduction is contradictory. Nevertheless, it has been suggested that MLD may also be effective in fibrotic tissue. However, although there are evaluation studies showing fibrosis in tissue with LE, there are no randomized controlled trials showing the effect of MLD and compression on fibrotic tissue in lower extremity LE. Similarly, there are no studies comparing the effect of lymphedema treatments on fibrosis using two different assessment methods. The primary aim of this study was to evaluate the effect of MLD applied as an adjunct to compression therapy on fibrosis in individuals with lower extremity LE. The secondary aim of the study was to evaluate the effect of MLD applied in addition to compression bandage on skin and subcutaneous tissue thickness, edema, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* According to the criteria of the International Society of Lymphology Stage 2 and 3 lower extremity LE to volunteer to participate in the study
* To be between the ages of 18-80
* LE involving the entire lower extremity

Exclusion Criteria:

* Acute deep vein thrombosis
* Acute infection
* Peripheral arterial disease in the lower extremity
* To have systemic diseases that may cause edema other than LE (renal failure, liver failure, heart failure, etc.)
* Chronic venous insufficiency
* Allergy to materials used in treatment
* Mental/cognitive problems that will affect cooperation
* Loss of sensation
* Presence of scleroderma in the treatment area
* Active cancer
* Radiogenic fibrosis in the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Fibrosis Using the SkinFibroMeter | Baseline, four week later and 3 month follow-up
  The patient will lie in a supine position on a treatment bed with the lower extremities relaxed. The SkinFibroMeter probe will be briefly (0.5 seconds) pressed perpendicularly against the skin. Each stiffness value will be calculated as the average of five consecutive successful measurements at the same site. If the applied force or measurement duration is incorrect, a 'USER ERROR' message will be displayed, and the measurements will be repeated.
  Fibrosis will be measured at 17 points on each lower extremity. Specific landmarks will be identified, including 5 cm above the joint of the second toe, 5 cm above the lateral malleolus, 10 cm below the inferior border of the patella, and 10 cm and 20 cm above the superior border of the patella. On the thigh and calf, medial, lateral, posterior, and anterior midline points corresponding to the same circumferential level as these landmarks will also be marked

SECONDARY OUTCOMES:
Assessment of Fibrosis Using Ultrasound | Baseline, four week later and 3 month follow-up
  The individual will lie in a supine position during the assessment. The thickness of the skin and subcutaneous tissue will first be measured without compression. Following this, maximum compression will be applied using an ultrasound probe to reassess the thickness for fibrosis evaluation. Maximum compression resistance is defined as the maximum pressure exerted to compress the tissue.
  Resistance to compression will be calculated in millimeters by subtracting the tissue thickness measured under maximum pressure from the initial thickness. This measurement will provide tissue compliance, enabling an indirect and objective assessment of fibrosis. A smaller difference indicates a higher propensity for fibrosis, while a larger difference suggests softer tissue.
  Fibrosis will be assessed at 17 points on each lower extremity.
Assessment of Skin and Subcutaneous Tissue Thickness | Baseline, four week later and 3 month follow-up
  The evaluation of skin and subcutaneous tissue thickness will be performed by a specialized radiologist using a LOGIQ ultrasound system (GE Healthcare, USA) equipped with a 6-15 MHz linear probe. Measurements will be conducted with the individual in a supine position. To optimize the passage of ultrasound waves, ultrasound gel will be applied between the probe and the skin. The ultrasound probe will be positioned perpendicularly to the skin, and brightness mode (B-mode) images will be obtained without applying additional compression to the skin. For skin thickness, the measurement will include the distance between two fine echogenic lines encompassing the hypoechoic dermis, as described comprehensively in previous studies, and will be recorded in millimeters. The subcutaneous distance will be measured as the distance in millimeters between the posterior echogenic line of the dermis and the anterior echogenic line of the muscular fascia
Edema Assessment | Baseline, four week later and 3 month follow-up
  Edema will be assessed by circumference measurements with the patient in a supine position. Measurements will start 10 cm from the heel. Along the lateral aspect of the leg, marks will be made at 8 cm intervals, and circumference measurements will be taken at these points along the extremity.
  Using a non-elastic tape measure 1 cm in width, measurements will be conducted without compressing the tissue and ensuring the ends of the tape do not overlap. Measurements will be recorded in centimeters. This process will be performed bilaterally.
  The recorded circumferences will then be converted into volume using the truncated cone formula, as extremities are considered geometrically as truncated cones for this calculation.
Assessment of Quality of Life | Baseline, four week later and 3 month follow-up
  The Lymphedema Quality of Life Questionnaire - Lower Limb (LYMQOL) will be used to assess quality of life. LYMQOL consists of 23 questions across four subdomains: function, mood, appearance, and symptoms. Each question is rated on a four-point Likert scale, where "1" indicates no impact and "4" indicates severe impact. The final question uses a numerical visual analog scale to evaluate overall quality of life.
  The questionnaire score is calculated by summing the scores of all questions and dividing by the total number of questions. The total score ranges from 1 to 4, with higher scores indicating worse quality of life. The Turkish validity and reliability of the questionnaire were established by Bakar et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zampell JC, Aschen S, Weitman ES, Yan A, Elhadad S, De Brot Andrade M, Mehrara BJ. Regulation of adipogenesis by lymphatic fluid stasis: part I. Adipogenesis, fibrosis, and inflammation. Plast Reconstr Surg. 2012 Apr;129(4):825-834. doi: 10.1097/PRS.0b013e3182450b2d. PMID 22456354
- [Background] Yamamoto T, Yamamoto N, Hayashi N, Hayashi A, Koshima I. Practicality of the Lower Extremity Lymphedema Index: Lymphedema Index Versus Volumetry-Based Evaluations for Body-Type-Corrected Lower Extremity Volume Evaluation. Ann Plast Surg. 2016 Jan;77(1):115-8. doi: 10.1097/SAP.0000000000000362. PMID 26835820
- [Background] Tashiro K, Feng J, Wu SH, Mashiko T, Kanayama K, Narushima M, Uda H, Miyamoto S, Koshima I, Yoshimura K. Pathological changes of adipose tissue in secondary lymphoedema. Br J Dermatol. 2017 Jul;177(1):158-167. doi: 10.1111/bjd.15238. Epub 2017 Apr 2. PMID 28000916
- [Background] Szuba A, Rockson SG. Lymphedema: classification, diagnosis and therapy. Vasc Med. 1998;3(2):145-56. doi: 10.1177/1358836X9800300209. PMID 9796078
- [Background] Szolnoky G, Dobozy A, Kemeny L. Towards an effective management of chronic lymphedema. Clin Dermatol. 2014 Sep-Oct;32(5):685-91. doi: 10.1016/j.clindermatol.2014.04.017. PMID 25160111
- [Background] Suehiro K, Morikage N, Murakami M, Yamashita O, Samura M, Hamano K. Significance of ultrasound examination of skin and subcutaneous tissue in secondary lower extremity lymphedema. Ann Vasc Dis. 2013;6(2):180-8. doi: 10.3400/avd.oa.12.00102. Epub 2013 May 10. PMID 23825499
- [Background] Reed JL, Pipe AL. The talk test: a useful tool for prescribing and monitoring exercise intensity. Curr Opin Cardiol. 2014 Sep;29(5):475-80. doi: 10.1097/HCO.0000000000000097. PMID 25010379
- [Background] Mosti G, Cavezzi A. Compression therapy in lymphedema: Between past and recent scientific data. Phlebology. 2019 Sep;34(8):515-522. doi: 10.1177/0268355518824524. Epub 2019 Jan 9. No abstract available. PMID 30626269
- [Background] Lim CY, Seo HG, Kim K, Chung SG, Seo KS. Measurement of lymphedema using ultrasonography with the compression method. Lymphology. 2011 Jun;44(2):72-81. PMID 21949976
- [Background] Li CY, Kataru RP, Mehrara BJ. Histopathologic Features of Lymphedema: A Molecular Review. Int J Mol Sci. 2020 Apr 6;21(7):2546. doi: 10.3390/ijms21072546. PMID 32268536
- [Background] Lee DG, Lee S, Kim KT. Computed Tomography-Based Quantitative Analysis of Fibrotic Changes in Skin and Subcutaneous Tissue in Lower Extremity Lymphedema Following Gynecologic Cancer Surgery. Lymphat Res Biol. 2022 Oct;20(5):488-495. doi: 10.1089/lrb.2021.0069. Epub 2022 Jan 10. PMID 35012367
- [Background] Leduc O, Leduc A, Bourgeois P, Belgrado JP. The physical treatment of upper limb edema. Cancer. 1998 Dec 15;83(12 Suppl American):2835-9. doi: 10.1002/(sici)1097-0142(19981215)83:12b+3.0.co;2-v. PMID 9874408
- [Background] Executive Committee. The Diagnosis and Treatment of Peripheral Lymphedema: 2016 Consensus Document of the International Society of Lymphology. Lymphology. 2016 Dec;49(4):170-84. PMID 29908550
- [Background] Brorson H. From lymph to fat: liposuction as a treatment for complete reduction of lymphedema. Int J Low Extrem Wounds. 2012 Mar;11(1):10-9. doi: 10.1177/1534734612438550. Epub 2012 Feb 23. PMID 22363050
- [Background] Bernas M, Thiadens SRJ, Stewart P, Granzow J. Secondary lymphedema from cancer therapy. Clin Exp Metastasis. 2022 Feb;39(1):239-247. doi: 10.1007/s10585-021-10096-w. Epub 2021 May 5. PMID 33950413
- [Background] Bakar Y, Tugral A. Translation, reliability, and validation of the Turkish version of the Lymphedema Quality-of-Life tool in Turkish-speaking patients with lower limb Lymphedema. J Vasc Nurs. 2019 Mar;37(1):11-17. doi: 10.1016/j.jvn.2018.11.005. Epub 2019 Jan 31. PMID 30954192
- [Background] Bakar Y, Ozdemir OC, Sevim S, Duygu E, Tugral A, Surmeli M. Intra-observer and inter-observer reliability of leg circumference measurement among six observers: a single blinded randomized trial. J Med Life. 2017 Jul-Sep;10(3):176-181. PMID 29075347
- [Background] Tzani I, Tsichlaki M, Zerva E, Papathanasiou G, Dimakakos E. Physiotherapeutic rehabilitation of lymphedema: state-of-the-art. Lymphology. 2018;51(1):1-12. PMID 30248726
- [Background] Sen EI, Arman S, Zure M, Yavuz H, Sindel D, Oral A. Manual Lymphatic Drainage May Not Have an Additional Effect on the Intensive Phase of Breast Cancer-Related Lymphedema: A Randomized Controlled Trial. Lymphat Res Biol. 2021 Apr;19(2):141-150. doi: 10.1089/lrb.2020.0049. Epub 2020 Oct 15. PMID 33058746
- [Background] Schaverien MV, Moeller JA, Cleveland SD. Nonoperative Treatment of Lymphedema. Semin Plast Surg. 2018 Feb;32(1):17-21. doi: 10.1055/s-0038-1635119. Epub 2018 Apr 9. PMID 29636649
- [Background] Rutkowski JM, Markhus CE, Gyenge CC, Alitalo K, Wiig H, Swartz MA. Dermal collagen and lipid deposition correlate with tissue swelling and hydraulic conductivity in murine primary lymphedema. Am J Pathol. 2010 Mar;176(3):1122-9. doi: 10.2353/ajpath.2010.090733. Epub 2010 Jan 28. PMID 20110415
- [Background] Lynch LL, Mendez U, Waller AB, Gillette AA, Guillory RJ 2nd, Goldman J. Fibrosis worsens chronic lymphedema in rodent tissues. Am J Physiol Heart Circ Physiol. 2015 May 15;308(10):H1229-36. doi: 10.1152/ajpheart.00527.2013. Epub 2015 Mar 13. PMID 25770241
- [Background] Ezzo J, Manheimer E, McNeely ML, Howell DM, Weiss R, Johansson KI, Bao T, Bily L, Tuppo CM, Williams AF, Karadibak D. Manual lymphatic drainage for lymphedema following breast cancer treatment. Cochrane Database Syst Rev. 2015 May 21;2015(5):CD003475. doi: 10.1002/14651858.CD003475.pub2. PMID 25994425
- [Background] Brouillard P, Witte MH, Erickson RP, Damstra RJ, Becker C, Quere I, Vikkula M. Primary lymphoedema. Nat Rev Dis Primers. 2021 Oct 21;7(1):77. doi: 10.1038/s41572-021-00309-7. PMID 34675250
- [Background] Azhar SH, Lim HY, Tan BK, Angeli V. The Unresolved Pathophysiology of Lymphedema. Front Physiol. 2020 Mar 17;11:137. doi: 10.3389/fphys.2020.00137. eCollection 2020. PMID 32256375
- [Background] Avraham T, Clavin NW, Daluvoy SV, Fernandez J, Soares MA, Cordeiro AP, Mehrara BJ. Fibrosis is a key inhibitor of lymphatic regeneration. Plast Reconstr Surg. 2009 Aug;124(2):438-450. doi: 10.1097/PRS.0b013e3181adcf4b. PMID 19644258
- [Background] Adriaenssens N, Belsack D, Buyl R, Ruggiero L, Breucq C, De Mey J, Lievens P, Lamote J. Ultrasound elastography as an objective diagnostic measurement tool for lymphoedema of the treated breast in breast cancer patients following breast conserving surgery and radiotherapy. Radiol Oncol. 2012 Dec;46(4):284-95. doi: 10.2478/v10019-012-0033-z. Epub 2012 Nov 9. PMID 23412910